CLINICAL TRIAL: NCT04798625
Title: A Norwegian Study of Vaccine Response to COVID-19 Vaccines in Patients Using Immunosuppressive Medication Within Rheumatology and Gastroenterology: the Nor-vaC Study
Brief Title: Vaccine Response to COVID-19 Vaccines in Patients Using Immunosuppressive Medication
Acronym: Nor-vaC
Status: Active, not recruiting | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Guro Løvik Goll, Principal investigator, Diakonhjemmet Hospital
Other Study IDs: DIA2021-1
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Spondyloarthritis; Crohn Disease; Ulcerative Colitis; Autoimmune Hepatitis; Liver Transplant; Complications
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis; Crohn Disease; Colitis, Ulcerative; Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum White blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Rheumatoid arthritis: Patients with a clinical diagnosis of rheumatoid arthritis and treated with immunosuppressive medication
- Psoriatic arthritis: Patients with a clinical diagnosis of psoriatic arthritis and treated with immunosuppressive medication
- Spondyloarthritis: Patients with a clinical diagnosis of spondyloarthritis and treated with immunosuppressive medication
- Crohn disease: Patients with a clinical diagnosis of Crohn disease and treated with immunosuppressive medication
- Ulcerative colitis: Patients with a clinical diagnosis of ulcerative colitis and treated with immunosuppressive medication
- Autoimmune hepatitis: Patients with a diagnosis of autoimmune hepatitis and treated with immunosuppressive medication
- Liver transplant: Patients who have undergone liver transplantation and are treated with immunosuppressive drugs

SUMMARY:
The purpose of this study is to assess the strength and duration of the immunological response to COVID-19 vaccines in patients treated with immunosuppressive and/or immunomodulating medication for immune-mediated inflammatory diseases in rheumatology and gastroenterology and after a liver transplantation.

DETAILED DESCRIPTION:
Patients on long-term immunosuppressive and/or immunomodulating medication may be susceptible to serious COVID-19. Hence, it is important they get sufficient protection by a COVID-19 vaccine. However, these patients may also be at risk for a less robust vaccine response. There is an urgent need to assess the humoral and cellular immune response to COVID-19 vaccines in these patient groups. The clinical consequences could be to administer several re-vaccinations or to adjust medication. This prospective, observational study aims to assess the immune response after COVID vaccination in patients suffering from inflammatory diseases and using immunosuppressive medication. Also, liver transplanted patients on immunosuppressive medication will be included.

Serum and whole blood samples will be obtained from all participants before and 1-4 weeks after the vaccination. Additionally, serum samples will be collected every 3-6 months for 5 years. If patients are allotted further vaccine doses , the patient response will be assessed by blood tests 2-4 weeks after any additional vaccine doses. In a subset of patients, samples will be drawn to study cellular immune responses. Demographic data and data regarding immunosuppressive medication will be recorded. Disease activity (clinical activity indices and biomarkers of inflammation) will be assessed. Blood samples will be obtained for biobank. Information regarding vaccination status and potential COVID-19 testing will be obtained from relevant registers.

ELIGIBILITY:
Inclusion Criteria:

1. An established clinical diagnosis of one of the following immune-mediated diseases: rheumatoid arthritis (RA), spondyloarthritis (SpA), psoriatic arthritis (PsA), ulcerative colitis (UC,) Crohns disease (CD), autoimmune hepatitis (AIH) or patients who have undergone a liver transplantation
2. Treatment with relevant immunosuppressive and/or immunomodulating medication *
3. Adult patients (> 18 years)
4. Patient intends to obtain vaccination against COVID-19 during the next 6 months

   * * The following drugs are considered relevant immunosuppressants and/or immunomodulators and patients using them may be eligible for this study: Rituximab, infliximab, adalimumab, golimumab, certolizumab, etanercept, tocilizumab, abatacept, secukinumab, vedolizumab, ustekinumab, risankizumab, methotrexate, sulfasalazine, leflunomide, azathioprine, 6-mercaptopurine, tofacitinib, filgotinib, baricitinib, upadacitinib, tacrolimus, mycophenolate, prednisolone

Exclusion Criteria:

1) Allergy or intolerance to elements of the COVID-19 vaccines

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidate patients will be recruited from the population treated at the two study centres and, if eligible, asked to participate in the observational cohort
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Serological response | 4 weeks after vaccination, then at 3 month intervals during the first year and 6 month intervals for up to a total of 5 years
  Change from baseline in serum levels of anti-SARS-CoV-2 antibodies

SECONDARY OUTCOMES:
Cellular response | 7-10 days after vaccination, then at 3 month intervals during the first year and 6 month intervals for up to a total of 5 years
  Change from baseline in T cell reactivity to SARS-CoV-2
Adverse events | Reported by patient for the first 48 hours following each vaccine dose
  Occurence of patient-reported adverse events related to vaccination against COVID-19
BASDAI | Within 4 weeks of the patient receiving the final dose of vaccine
  BASDAI questionnaire to assess disease activity in spondyloarthritis
Partial Mayo score | Every 3 months for the first year of study, every 6 months thereafter until study completion
  Partial Mayo score to assess disease activity in ulcerative colitis
Harvey-Bradshaw index (HBI) | Every 3 months for the first year of study, every 6 months thereafter until study completion
  Harvey-Bradshaw index to assess disease activity in Crohn disease
DAS28 | Within 4 weeks of the patient receiving the final dose of vaccine
  Disease Activity Score 28 to assess disease activity in RA and PsA

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Diakonhjemmet Hospital, Oslo

REFERENCES:
- [Result] Jyssum I, Kared H, Tran TT, Tveter AT, Provan SA, Sexton J, Jorgensen KK, Jahnsen J, Kro GB, Warren DJ, Vaage EB, Kvien TK, Nissen-Meyer LH, Anderson AM, Grodeland G, Haavardsholm EA, Vaage JT, Mjaaland S, Syversen SW, Lund-Johansen F, Munthe LA, Goll GL. Humoral and cellular immune responses to two and three doses of SARS-CoV-2 vaccines in rituximab-treated patients with rheumatoid arthritis: a prospective, cohort study. Lancet Rheumatol. 2022 Mar;4(3):e177-e187. doi: 10.1016/S2665-9913(21)00394-5. Epub 2021 Dec 23. PMID 34977602
- [Result] Syversen SW, Jyssum I, Tveter AT, Tran TT, Sexton J, Provan SA, Mjaaland S, Warren DJ, Kvien TK, Grodeland G, Nissen-Meyer LSH, Ricanek P, Chopra A, Andersson AM, Kro GB, Jahnsen J, Munthe LA, Haavardsholm EA, Vaage JT, Lund-Johansen F, Jorgensen KK, Goll GL. Immunogenicity and Safety of Standard and Third-Dose SARS-CoV-2 Vaccination in Patients Receiving Immunosuppressive Therapy. Arthritis Rheumatol. 2022 Aug;74(8):1321-1332. doi: 10.1002/art.42153. Epub 2022 Jun 29. PMID 35507355
- [Result] Christensen IE, Jyssum I, Tveter AT, Sexton J, Tran TT, Mjaaland S, Kro GB, Kvien TK, Warren DJ, Jahnsen J, Munthe LA, Haavardsholm EA, Vaage JT, Grodeland G, Lund-Johansen F, Jorgensen KK, Syversen SW, Goll GL, Provan SA. The persistence of anti-Spike antibodies following two SARS-CoV-2 vaccine doses in patients on immunosuppressive therapy compared to healthy controls-a prospective cohort study. BMC Med. 2022 Oct 5;20(1):378. doi: 10.1186/s12916-022-02587-8. PMID 36199139
- [Result] Syversen SW, Jyssum I, Tveter AT, Sexton J, Christensen IE, Tran TT, Bjorlykke KH, Mjaaland S, Warren DJ, Kvien TK, Chopra A, Kro GB, Jahnsen J, Munthe LA, Haavardsholm EA, Grodeland G, Vaage JT, Provan SA, Jorgensen KK, Goll GL. Immunogenicity and safety of a three-dose SARS-CoV-2 vaccination strategy in patients with immune-mediated inflammatory diseases on immunosuppressive therapy. RMD Open. 2022 Nov;8(2):e002417. doi: 10.1136/rmdopen-2022-002417. PMID 36328399
- [Result] Bjorlykke KH, Orbo HS, Tveter AT, Jyssum I, Sexton J, Tran TT, Christensen IE, Kro GB, Kvien TK, Jahnsen J, Munthe LA, Chopra A, Warren DJ, Mjaaland S, Haavardsholm EA, Grodeland G, Provan SA, Vaage JT, Syversen SW, Goll GL, Jorgensen KK. Four SARS-CoV-2 vaccine doses or hybrid immunity in patients on immunosuppressive therapies: a Norwegian cohort study. Lancet Rheumatol. 2023 Jan;5(1):e36-e46. doi: 10.1016/S2665-9913(22)00330-7. Epub 2022 Nov 16. PMID 36415604
- [Result] Jorgensen KK, Hoivik ML, Chopra A, Benth JS, Ricanek P, Moum PB, Jyssum I, Bolstad N, Warren DJ, Vaage PJT, Munthe PLA, Lundin PKEA, Anisdahl K, Syversen SW, Goll GL, Lund-Johansen F, Medhus AW, Jahnsen PJ. Humoral immune response to SARS-CoV-2 vaccination in patients with inflammatory bowel disease on immunosuppressive medication: association to serum drug levels and disease type. Scand J Gastroenterol. 2023 Jul-Dec;58(8):874-882. doi: 10.1080/00365521.2023.2177884. Epub 2023 Feb 14. PMID 36788656
- [Derived] Orbo HS, Bjorlykke KH, Sexton J, Jyssum I, Tveter AT, Christensen IE, Mjaaland S, Kvien TK, Grodeland G, Kro GB, Jahnsen J, Haavardsholm EA, Munthe LA, Provan SA, Vaage JT, Goll GL, Jorgensen KK, Syversen SW. Incidence and outcome of COVID-19 following vaccine and hybrid immunity in patients on immunosuppressive therapy: identification of protective post-immunisation anti-RBD antibody levels in a prospective cohort study. RMD Open. 2024 Apr 9;10(2):e003545. doi: 10.1136/rmdopen-2023-003545. PMID 38599653